CLINICAL TRIAL: NCT01355367
Title: A Multicenter, Open Label, Long Term Extension Study of Oral BAYA1040 CR 80 mg (40 mg Bid) for 44 Weeks in Patients With Essential Hypertension (Extension From Study 13176)
Brief Title: High Dose BAYA1040 CR: a Long Term Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14023
Record Dates: First submitted 2011-04-21; First posted 2011-05-18 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: BAYA1040 CR; Nifedipine; Essential hypertension; Japanese Patients; Phase III; Extension study
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Nifedipine (Adalat, BAYA1040)

INTERVENTIONS:
Drug: Nifedipine (Adalat, BAYA1040) — BAYA1040 CR 40mg BID

SUMMARY:
This is a clinical study evaluating the safety and efficacy of long term administration of oral BAYA1040 CR 80 mg/day (40 mg twice daily) in patients with essential hypertension for whom the test drug is tolerable during the 8 week double blind treatment phase of Study 13176.

ELIGIBILITY:
Inclusion Criteria:

* Patients who complete the 8 week double blind treatment phase of Study 13176 and for whom the test drug is tolerable

Exclusion Criteria:

* Patients with expected difficulties for the continuous 1 year follow up

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events collection | Week 52

SECONDARY OUTCOMES:
Changes from baseline in diastolic blood pressure (DBP) while sitting | Baseline, week 10, 12, 16, 24, 28, 32, 36, 40, 44, 48 and 52
Changes from baseline in systolic blood pressure (SBP) while sitting | Baseline, week 10, 12, 16, 24, 28, 32, 36, 40, 44, 48 and 52
Proportion of subjects achieving a target BP based on the Japanese Society of Hypertension (JSH) 2009 guidelines | Baseline, week 10, 12, 16, 24, 28, 32, 36, 40, 44, 48 and 52
Proportion of subjects achieving a target DBP and SBP based on JSH 2009 guidelines or a >10 mmHg reduction of DBP | Baseline, week 10, 12, 16, 24, 28, 32, 36, 40, 44, 48 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Japan (13):
  - Hirosaki, Aomori
  - Kamagaya, Chiba
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Kawasaki, Kanagawa
  - Daitō, Osaka
  - Kishiwada, Osaka
  - Yao, Osaka
  - Tokorozawa, Saitama
  - Shizuoka, Shizuoka
  - Hachiōji, Tokyo
  - Meguro City, Tokyo
  - Minato, Tokyo